CLINICAL TRIAL: NCT04929470
Title: Clinical Investigation of the Safety and Performance of HiResTM Ultra Cl HiFocusTM SlimJ Electrode (Cl-1600-05) and HiResTM Ultra 3D Cl HiFocusTM SlimJ Electrode (Cl-1601-05) (Ultra X) in Adults With Severe-to-profound Hearing Loss
Brief Title: Safety and Performance of Ultra/Ultra 3D Cl With HiFocus SlimJ Electrode in Adults With Severe-to-profound Hearing Loss
Status: Active, not recruiting | Type: Observational
Sponsor: Advanced Bionics AG (Industry)
Responsible Party: Sponsor
Other Study IDs: ABIntl-19-45
Record Dates: First submitted 2021-06-06; First posted 2021-06-18 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Cochlear Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — Cochlear Implantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: cochlear implantation — patients receive a cochlear implantation within clinical routine

SUMMARY:
This is a prospective study designed to evaluate the safety and performance of the HiResTM Ultra Cl HiFocusTM SlimJ Electrode and HiResTM Ultra 3D Cl HiFocusTM SlimJ Electrode (Ultra X) under normal conditions of use as it is approved for this device. Participants receive interventions as part of routine medical care.

DETAILED DESCRIPTION:
This study is set up to document any adverse events and comparing pre- to post-implant benefit to subjects. Any adverse events associated with the device will be documented via Advanced Bionics complaint handling system for the lifetime of the device. A within-subjects repeated-measures design will be employed. Speech perception will be evaluated preoperatively with conventional amplification to determine candidacy and to establish baseline performance. Efficacy parameters are speech perception data which will be collected according to clinical routine with a 6 month follow up period. Subjects will be implanted unilaterally with the Ultra X according to standard clinical care.

The primary efficacy objective is to demonstrate that mean monosyllabic word recognition score with the Ultra X used in combination with a sound processor programmed with the latest fitting software six months after activation is at least 20% better than the mean word score at baseline with conventional amplification in the same ear.

The primary efficacy endpoint is reached six months after device activation.

ELIGIBILITY:
Inclusion Criteria:

* No previous experience with any auditory implant
* 18 years of age or older
* Postlingual onset of severe hearing loss (≥ 4 years of age)
* Limited benefit from appropriately fitted hearing aids, defined as scoring 60% or less in Freiburger Monosyllabic word test
* German language proficiency
* Willingness to participate in all scheduled procedures outlined in the protocol

Exclusion Criteria:

* Cochlear malformation or obstruction that would preclude full insertion of electrode array.
* Presence of additional disabilities that would prevent or interfere with participation in the required study procedures
* Medical or psychological conditions that contraindicate surgery or impact the ability to manage an implanted device or the study related procedures
* Evidence of central auditory lesion or compromised auditory nerve
* Pregnancy at time of surgery.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 30 adult subjects with valid and useable data
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-07-06 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Speech recognition score (word score) | 6 months
  The primary efficacy objective is to demonstrate that mean monosyllabic word recognition score (Minimum Score 0 percent and maximum score 100 percent wheras 0 percent is worse and 100 is better) with the Ultra implants used in combination with a sound processor programmed with the latest fitting software is at least 20 percent better than the mean monosyllabic word score at baseline with conventional amplification in the same ear.
Analysis of participants with device failure | 6 months
  A maximum of one device failure that require device replacement during the first six months following device activation (activation approximately one to eight weeks after surgery).

SECONDARY OUTCOMES:
Analysis of Speech reception threshold | 6 months
  50 percent speech reception threshold in the Oldenburger Sentence Test (OlSa) in noise in the implanted ear six months after device activation compared to baseline performance with conventional amplification in the same ear.

OTHER OUTCOMES:
Device fitting data | 6 months
  M-level [CU] CU=Clinical Units
Device verification data | 6 months
  Impedances [Kilo Ohm]
Professional feedback from the audiologist using the latest fitting software to program the latest processor | 6 months
  Feedback will be collected with a structured questionnaire
Feedback from the surgeon on handling of the device and tools during implantation | 6 months
  Feedback will be collected with a structured questionnaire
hours of usage | 6 months
  hours of usage as summarized in the logging of the processor
using habits of participants | 6 months
  Assessement with a structured patient questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Arneborg Ernst, Prof. Dr., Principal Investigator — Unfallkrankenhaus Berlin
Locations (3):
- Germany (3):
  - HNO-Klinik Düsseldorf, Düsseldorf, Düsseldorf
  - Unfallkrankenhaus Berlin (UKB), Berlin, State of Berlin
  - Westfälische Wilhelms-Universität Münster, Münster

IPD SHARING:
Plan to Share IPD: Undecided